CLINICAL TRIAL: NCT02641964
Title: Risk Factors for ARDS in Patients With Acute Necrotizing Pancreatitis
Status: Completed | Type: Observational
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Bin He, Emergency department physician, Nanjing Medical University
Other Study IDs: JSSRMYY-HB-1
Record Dates: First submitted 2015-12-08; First posted 2015-12-30 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Acute Necrotizing Pancreatitis; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ARDS group: patients with acute necrotizing pancreatitis complicated by ARDS
- non-ARDS group: acute necrotizing pancreatitis patients without ARDS

SUMMARY:
Try to collect about 350 cases of acute necrotizing pancreatitis at the First Affiliated Hospital with Nanjing Medical University and Nanjing General Hospital of Nanjing Military Command. Then the investigators studied the incidence and the risk factors of ARDS in patients with acute necrotizing pancreatitis.

DETAILED DESCRIPTION:
Using electronic patient data monitoring systems, the investigators reviewed all patients with a diagnosis of pancreatitis admitted to surgical wards or ICUs at the First Affiliated Hospital with Nanjing Medical University and Nanjing General Hospital of Nanjing Military Command from January 1, 2009, to October 31, 2015. Inclusion criteria were adult patients (age >18 years) with acute necrotizing pancreatitis. Exclusion criteria were as follows : 1) lack of radiologic evidence to diagnose acute necrotizing pancreatitis, 2) presence of ARDS before admission to hospitals, 3) unable to partner treatment and leaving hospitals, 4) transferring to the investigators' hospitals after treatment, 5) missing other necessary data, and 6) pregnancy.

For enrolled patients, general clinical characteristics were collected. Patients were categorized into two groups according to ARDS or non-ARDS, and the differences of these characteristics between two groups were evaluated. Potential risk factors were collected and studied by using multiple logistic regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age >18 years) with acute necrotizing pancreatitis

Exclusion Criteria:

* lack of radiologic evidence to diagnose acute necrotizing pancreatitis,
* presence of ARDS before admission to hospitals,
* unable to partner treatment and leaving hospitals,
* transferring to the investigators' hospitals after treatment,
* missing other necessary data,
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the investigators reviewed all patients with a diagnosis of pancreatitis admitted to surgical wards or ICUs at the First Affiliated Hospital with Nanjing Medical University and Nanjing General Hospital of Nanjing Military Command from January 1, 2009, to October 31, 2015.Adult patients (age >18 years) with acute necrotizing pancreatitis were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2015-11; Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
the incidence of ARDS in patients with acute necrotizing pancreatitis | up to 2 months

SECONDARY OUTCOMES:
the risk factors for ARDS in patients with acute necrotizing pancreatitis | up to 2 months
  Potential risk factors included smoking, alcohol abuse, diabetes mellitus, abdominal surgery, shock, hypoalbuminaemia, hypertriglyceridemia and hypercholesterolemia.Univariate analyses examined potential risk factors on outcome (ARDS or non-ARDS). Then, using multiple logistic regression analysis, factors achieving P≤0.1 in univariate analyses were entered into the model predicting the risk for the onset of ARDS.

OTHER OUTCOMES:
the effect of ARDS on mortality in patients with severe acute pancreatitis | up to 2 months
  The mortality were compared between ARDS and non-ARDS patients with severe acute pancreatitis. The differences were evaluated by χ2 or Fisher exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Bin He, Master, Study Director — Nanjing Medical University

IPD SHARING:
Plan to Share IPD: Yes